CLINICAL TRIAL: NCT04381091
Title: Expanded Access Program for Idebenone in Patients With Leber's Hereditary Optic Neuropathy Who Completed the LEROS Study
Acronym: US EAP LHON
Status: No longer available | Type: Expanded Access
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: SNT-EAP-IDE-004
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Leber's Hereditary Optic Neuropathy
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber | interventions — idebenone; Tablets

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Idebenone 150 MG Oral Tablet — idebenone 900 mg/day

SUMMARY:
Expanded Access Program for Idebenone in Patients with Leber's Hereditary Optic Neuropathy who completed the LEROS Study

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the LEROS study, who attended the end of study visit in LEROS and who in the opinion of investigator could benefit from continuation of idebenone treatment.
* Signed and dated Informed Consent Form (to be obtained at the Enrollment Visit from patient or parent/legal guardian (if applicable) prior to dispensing idebenone to the patient).

Exclusion Criteria:

* Patients who, in the opinion of the LEROS investigator, had unacceptable tolerability of idebenone treatment in LEROS trial.
* Patients who prematurely discontinued the LEROS study.

Sex: All
Age Groups: Child, Adult, Older Adult